CLINICAL TRIAL: NCT03916575
Title: National Multicenter Retrospective Study: PEComas: Natural History and Prognostic
Brief Title: PEComas: Natural History and Prognostic Factors
Acronym: PEComas
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7337
Record Dates: First submitted 2019-04-03; First posted 2019-04-16 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: PEComas
MeSH Terms: conditions — Perivascular Epithelioid Cell Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Perivascular epithelioid cell tumors are rare and characterized by the expression of myomelanocytic markers. They belong to a complex tumor family that includes angiomyolipomas, lymphangioleiomyomatosis and other soft-tissue tumors. Given their rarity, the natural history of pecomas is not yet understood, and a comprehensive classification that integrates clinical, pathological and molecular features has not been achieved as of today.

This study is a national multicenter retrospective study to better understand the natural history of PEComas, excluding lymphangioleiomyomatosis and classic triphasic angiomyolipomas.

The primary purpose is the identification of prognostic markers impacting the relapse. Secondaries purposes are to identify prognostic markers impacting the overall survival and to have a better understanding of natural history

ELIGIBILITY:
Inclusion Criteria:

* Major patient (≥18 years old)
* Minor patient (1 to 17 years old)
* PEComas diagnosed in France between 1990 and 2018 and read back by a pathologist referent of sarcomas
* Patient having agreed to the use of his medical data for the purpose of this research.
* Parental authorities having given their agreement for the reuse of their child's medical data for the purpose of this research.

Exclusion Criteria:

* Opposition of the patient (or his legal representative) to the reuse of his data for the purposes of this research
* Impossibility of giving the subject clear information
* Patient under safeguard of justice
* Patient under guardianship
* Lymphangioleiomyomatosis
* Classic triphasic angiomyolipoma

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient having PEComas diagnosed in France between 1990 and 2018
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-04-09 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Study of the prognostic factors associated with the risk of relapse | The period from January 1st, 1990 to December 31, 2018 will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Service D'Hematologie Et D'Oncologie, Strasbourg, France